CLINICAL TRIAL: NCT03820128
Title: Very Early and Early Nutrition in Acute Pancreatitis in Children: a Randomized Study
Brief Title: Early Nutrition in Acute Pancreatitis
Acronym: OZT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OZT
Record Dates: First submitted 2018-06-14; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-06

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very early refeeding (Active Comparator): Very early diet intervention: refeeding within 24 hours from the hospital admission.
  Participants will be encouraged to start eating immediately after the time of admission. They will be able to choose the meal from the list with no amount or calories restriction.They will be asked to conduct the daily diet diary - time of feeding, quality and quantity of the foods ingested. Laboratory tests will be performed at the study entry, on the day of 3 and 5 of hospitalization and on the day of discharge.
  Interventions: Other: Early diet intervention
- Early refeeding (Active Comparator): Early diet intervention: refeeding after 24 hours from the hospital admission .
  During the first 24 hours after admission participants will be on fluid only (orally and/or intravenously). Later on they will be encouraged to start eating. They will be able to choose the meal from the list with no amount or calories restriction.They will be asked to conduct the daily diet diary - time of feeding, quality and quantity of the foods ingested. Laboratory tests will be performed at the study entry, on the day of 3 and 5 of hospitalization and on the day of discharge.
  Interventions: Other: Early diet intervention

INTERVENTIONS:
Other: Early diet intervention — Participant's diet includes several low-fiber and low-fat commonly available meals and products. Patients will choose what they want to eat with no amount or calories restriction.

SUMMARY:
The aim of the study is to assess the effect of the early oral refeeding and fat content in the diet on the length of stay, clinical course (included pain severity) in pediatric patients with mild and moderate AP. Patients will be randomized to groups: refeeding within 24 hours or after 24 hours from the hospital admission. Biochemical tests and pain severity will be evaluated.

DETAILED DESCRIPTION:
Prospective, randomized study. Research in the adult population shows that early enteral feeding in acute pancreatitis (AP) both oral and via the feeding tube is safe, shortens the length of hospital stay, prevents the multi organ failure (MoF) and reduces mortality. The pediatric population lacks prospective data concerning refeeding modes in AP. The aim of the study is to assess the effect of the early oral refeeding and fat content in the diet on the length of stay, clinical course (included pain severity) in pediatric patients with mild and moderate AP. Patients will be randomized to groups: refeeding within 24 hours or after 24 hours from the hospital admission. Biochemical tests including CRP, amylase, lipase and proinflammatory cytokines levels and zonulin level as well as severity of pain will be assessed again in the second, the third and the fifth hospital day.

ELIGIBILITY:
Inclusion Criteria:

* AP diagnosis according to the generally accepted criteria ie. fulfilling two out of three criteria:

  * Abdominal pain of pancreatic origin
  * Radiologic findings supportive of AP on imaging
  * Amylase or lipase levels elevation three times above the upper limit of normal
* Mild or moderate AP Mild AP: AP without organ failure, local or general complications Moderate AP: AP that may be accompanied by intermittent organ failure, local complications or concomitant disease worsening
* No contradictions to enteral treatment
* Informed consent from the parents or legal guardian and from the patient if older than 16 years

Exclusion Criteria:

* Severe general condition
* Severe AP
* Kidney insufficiency, cardiac insufficiency
* Diabetes type 1
* Cystic fibrosis
* Contraindications to enteral feeding
* Lack of required informed consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospitalization | through study completion, an average of 2 years
  Number days of hospitalization

SECONDARY OUTCOMES:
Time between the onset of symptoms and the first feeding | assessed at the day of 2
  Time between the onset of symptoms and the first feeding measured in hours
Adverse events | daily assessment in the first three days of hospitalization
  Severity of abdominal pain daily using a 10 point visual - analog scale (VAS). 0 means lack of the pain, 10 means the most severe pain
Average calories intake | through study completion, an average of 2 years
  Average calories intake (kcal)
Levels of proinflammatory cytokine levels. | through study completion, an average of 2 years
  Proinflammatory cytokine levels (ng/ml) using ELISA tests
Zonulin level | through study completion, an average of 2 years
  Zonulin level (ng/ml) using ELISA test

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Paediatric Gastroenterology and Nutrition., Warsaw, Poland